CLINICAL TRIAL: NCT06648213
Title: Investigation of the Effect of Individual Structured Therapy Application on Motor Performance in Early Premature Infants Hospitalized in Neonatal Intensive Care Unit
Brief Title: Individual Structured Therapy in Early Premature Infants at the Neonatal Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Özge ÇANKAYA, PT, PhD, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SBUNICU
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Infant Development; Neonatal Intensive Care Unit; INDIVIDUALIZED THERAPY
Keywords: individualized therapy, infant development, neonatal intensive care unit, early preterm
MeSH Terms: conditions — Premature Birth | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized Physiotherapy (Other): Therapy group: In addition to routine care, they will be arranged according to the needs of the baby in the form of positioning, hand contacts, passive and active movement of the arms and legs for the development of movement, sensory stimuli around the mouth for oral motor organisation. Neurodevelopmental-based application will be applied three days a week, once a day for 10-15 minutes, from the 34th week until 36th week when vital signs are stable.
  Interventions: Other: Physiotherapy
- Control (No Intervention): Control group: They will be monitored by performing routine care and positioning.

INTERVENTIONS:
Other: Physiotherapy — Therapy group: In addition to routine care, they will be arranged according to the needs of the baby in the form of positioning, hand contacts, passive and active movement of the arms and legs for the development of movement, sensory stimuli around the mouth for oral motor organisation. Neurodevelopmental-based application will be applied three days a week, once a day for 10-15 minutes, from the 34th week until 36th week when vital signs are stable.
  Arms: Individualized Physiotherapy

SUMMARY:
In this study, investigators aimed to apply an individual structured therapy protocol within the framework of neurodevelopmental therapy principles in early premature infants hospitalized in the neonatal intensive care unit and to examine its effect on the motor development of infants.

DETAILED DESCRIPTION:
The study is planned to include 20 early premature (<34 weeks) newborns hospitalised in the neonatal intensive care unit. The babies will be divided into two groups as therapy group and control group. Internet-based randomisation system will be used to determine the groups according to their risk levels. The risk levels will be determined according to the guidelines of the Turkish Neonatology Association.

Sterile gowns, masks and bonnets will be used during assessment and therapy to reduce the risk of infection in terms of the safety of the babies, and small lids will be opened so that the physiotherapist's hand can enter to maintain the temperature and oxygen balance in the incubator.

Therapy group: In addition to routine care, they will be arranged according to the needs of the baby in the form of positioning, hand contacts, passive and active movement of the arms and legs for the development of movement, sensory stimuli around the mouth for oral motor organisation. Neurodevelopmental-based application will be applied three days a week, once a day for 10-15 minutes, from the 34th week until 37th week when vital signs are stable.

Control group: They will be monitored by performing routine care and positioning.

ELIGIBILITY:
Inclusion criteria

1. Hospitalised in the neonatal intensive care unit,
2. Born before 34 weeks of gestation
3. medium and low-risk babies
4. Newborns who were approved by their families to participate in the study Exclusion criteria

1. Diagnosed neurological, neuromuscular or genetic disease 2. Congenital anomalies 3. Newborns whose parents did not consent to participate in the study

Max Age: 34 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
General Movements | For GMA analysis in our study, a 3-5 min video of the babies lying supine outside the incubator will be taken. The videos will be recorded at 34th week and 36th week.
  GMs movements are a complex set of movements involving the whole body of the baby, which start to be observed from the 9th week of intrauterine life, change shape after the second month of the postterm period and can be monitored until the 20th week in corrected form.
  GMA is a valid and reliable analysis used to determine brain dysfunctions in preterm, term and postterm infants up to the 20th week.
  GMA analysis can be performed during sleep or wakefulness in preterm infants.
Hammersmith Neonatal Neurological Examination (HNNE) | The HNNE short form will be applied at 34th week and 36th week.
  HNNE is a rapid, practical and easy-to-apply assessment method. It can be used in the assessment of term and preterm babies of different ages within the neonatal period. It is one of the standard methods used to predict the risk of cerebral palsy.

SECONDARY OUTCOMES:
Weigh | Three times a week between 34-36th weeks.
  Weight gain will be analyzed by recording daily weight.

CONTACTS AND LOCATIONS:
Locations (1):
- Gülhane Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided